CLINICAL TRIAL: NCT05458726
Title: Research on the Correlation Between Efficacy of Osimertinib and EGFR T790M Status and Ratio Via Digital Droplet PCR (ddPCR) From Peripheral Blood in NSCLC Patients
Brief Title: Correlation Between Efficacy of Osimertinib and EGFR T790M Status and Ratio Via ddPCR in NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Junling Li, Professor, Peking Union Medical College
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: NCC-005374
Record Dates: First submitted 2022-07-07; First posted 2022-07-14 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: EGFR T790M; Osimertinib; Non-small Cell Lung Cancer; ddPCR
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib; Paclitaxel; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Osimertinib (Experimental): Osimertinib 80mg po daily
  Interventions: Drug: Osimertinib
- Other treatments (Sham Comparator): chemotherapy or continuation of TKI monotherapy or in combination of anti-angiogenic agents
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — Osimertinib or chemotherapy
  Other Names: paclitaxel; carboplatin; pemetrexed

SUMMARY:
Liquid biopsy is emerging as an essential tool in tumor monitoring and a potential alternative and supplement to tissue biopsy for tumor genotyping, especially in relapsed or metastatic diseases. Liquid biopsy methods for detecting T790M in ctDNA can be qualitative or quantitative, including amplification refractory mutation system PCR (ARMS-PCR), digital droplet polymerase chain reaction (ddPCR), and next generation sequencing (NGS)-based methods. Comparison of multiple detecting platform for EGFR mutations in plasma samples has been undertaken in studies to determine the most feasible assay in clinical practice. In this study, we will investigate the usefulness of ddPCR for quantitative detection of EGFR T790M mutation in peripheral blood, and compared the utility of ddPCR and NGS for guiding decisions regarding osimertinib therapy in NSCLC patients who had develop resistance to first- or second generation EGFR-TKIs.

ELIGIBILITY:
Inclusion Criteria:

* histologically/cytologically confirmed stage IV NSCLC patients harboring sensitizing EGFR mutations;
* progression from first or second-generation EGFR-TKI confirmed by radiographic imaging;
* received both NGS test and ddPCR from peripheral blood simultaneously.

Exclusion Criteria:

* progression from first- or second-generation EGFR-TKIs as adjuvant therapy;
* having received third-generation EGFR-TKIs prior to the gene tests;
* having received NGS test only or ddPCR test only.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 1 year
  Time from initiation of osimertinib or other anti-tumor treatment to progression or death from any cause

SECONDARY OUTCOMES:
ORR | up to 1 year
  the sum of CR and PR rates
DCR | up to 1 year
  the sum of CR ,PR and SD rates

CONTACTS AND LOCATIONS:
Overall Officials: Junling Li, Professor, Principal Investigator — Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Junling Li, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu Z, Li Y, Wang L, Hao X, Ying J, Li J, Xing P. Efficacy of third-generation epidermal growth factor receptor-tyrosine kinase inhibitors in advanced NSCLC with different T790M statuses tested via digital droplet polymerase chain reaction ddPCR and next-generation sequencing. Expert Rev Anticancer Ther. 2024 Mar-Apr;24(3-4):183-192. doi: 10.1080/14737140.2024.2334807. Epub 2024 Apr 17. PMID 38526910